CLINICAL TRIAL: NCT03905720
Title: Non-pharmacologic Approaches to Relieve Pain and Symptom Distress Among Diverse Hospitalized Cancer Patients
Brief Title: Pragmatic Research of Acupuncture and Counseling eXtended to Inpatient Services
Acronym: PRACXIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-23446; NCI-2018-02204 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 18801 (Other: University of California, San Francisco)
Record Dates: First submitted 2018-08-30; First posted 2019-04-05 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Malignant Solid Tumor; Pain
Keywords: cancer; inpatient; non-pharmacologic approaches; pain management; acupuncture; pain counseling
MeSH Terms: conditions — Pain; Neoplasms; Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: 2x2 randomized factorial design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment As Usual (No Intervention): Participants will receive routine care consisting of usual analgesic medications for pain in adults with cancer.
- Acupuncture (Active Comparator): Along with routine pain medications, participants will be offered daily acupuncture treatments for up to four days.
  Interventions: Procedure: Acupuncture
- Pain Counseling (Active Comparator): Along with routine pain medications, participants will receive evidence-based psychosocial support through education and counseling provided by qualified study staff.
  Interventions: Behavioral: Pain Counseling
- Acupuncture and Pain Counseling (Active Comparator): Along with routine pain medications, participants will be offered daily acupuncture treatments and pain counseling for up to four days as described above.
  Interventions: Procedure: Acupuncture; Behavioral: Pain Counseling

INTERVENTIONS:
Procedure: Acupuncture — A licensed acupuncturist will assess participants' symptoms and administer acupuncture needles in accordance with traditional Chinese medicine principles and the study protocol. Treatments will provided daily for up to four hospital days.
  Arms: Acupuncture; Acupuncture and Pain Counseling
Behavioral: Pain Counseling — Participants will receive sessions with a counselor trained in pain management. The pain counselor will explain, review, and discuss the contents of a Pain Control booklet. Sessions will include pain assessment, pain education, and coping skills, provided daily for up to four hospital days.
  Arms: Acupuncture and Pain Counseling; Pain Counseling

SUMMARY:
Despite improved assessment and pharmacologic management, cancer pain is still undertreated. Using non-pharmacologic treatments alongside medications may better address patients' total pain experience by relieving physical and psychological symptoms and reducing the adverse effects of drugs. However, our knowledge of the benefits of multidisciplinary approaches in real-world hospital settings is limited. Patients want to know "How can I get the most pain relief with the fewest side effects?" This study proposal is designed to address this question by testing how combining pharmacologic and non-pharmacologic (acupuncture and pain counseling) treatments can: (1) maximize effectiveness, (2) minimize harms, and (3) align with patients' preferences.

DETAILED DESCRIPTION:
This study compares clinically-relevant therapeutic options in two high-volume hospitals (one public, one university) to address the core research question of whether non-pharmacologic approaches improve symptom management among diverse inpatients. Study investigators will assess the effectiveness of acupuncture and of pain counseling independently and in combination.

Participants will be randomized to two factors each with two levels, yielding four experimental conditions: (1) standard pharmacologic pain management, (2) pharmacologic pain management + acupuncture, (3) pharmacologic pain management + pain counseling, (4) pharmacologic pain management + acupuncture + pain counseling. Patient outcomes will be assessed using a mixed-methods approach, with validated scales for quantitative measures and qualitative interviews to elicit stakeholder perspectives (patients, caregivers, providers).

The study will be conducted as a pragmatic clinical trial at two hospitals to address these aims:

1. Determine the effectiveness of adjunctive acupuncture and of pain counseling for improving pain management.
2. Determine the extent that adjunctive acupuncture and pain counseling reduce use of opioid analgesics and side effects.
3. Examine stakeholder perspectives on non-pharmacologic approaches to pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to University of California San Francisco (UCSF) or Zuckerberg San Francisco General (ZSFG) with a malignant solid tumor
2. Speak Cantonese, English, or Spanish
3. Have an anticipated stay of ≥ 48 hours
4. Be aged 21 or older
5. Have pain intensity of ≥ 4 out of 10 for worst pain in the prior 24 hours when enrolled

Exclusion Criteria:

1. Acupuncture contraindication
2. Unstable medical condition (e.g., severe pulmonary disease, myocardial infarction)
3. Admission to the psychiatric ward (e.g., for severe depression)
4. Inability to consent (e.g., cognitive impairment)
5. Prior involvement with the study (e.g., readmissions)
6. Platelets < 50,000 microliters
7. Absolute neutrophil count < 500 microliters
8. C. difficile infection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in worst pain intensity assessed by the NRS | Daily for up to four hospital days
  Participants' worst level of pain in the past 24 hours on a 0-10 numeric rating scale (NRS), 0= no pain and 10= worst pain imaginable

SECONDARY OUTCOMES:
Use of opioids during hospital stay | Hospital stay (average length of stay = 5 days)
  Total and average daily use of opioids based on morphine milligram equivalence
Presence and severity of common side effects | Daily for up to four hospital days
  Nausea, vomiting, agitation, and sedation
Cancer-related distress | Daily for up to four hospital days
  Single item measure developed by the National Comprehensive Cancer Network. Participants are asked to indicate the number that best describes how much distress they are experiencing in the past week including today, 0=no distress and 10=extreme distress.
Health-related quality of life assessed by the EuroQol EQ-5D-3L (EQ-5D-3L) | Daily for up to four hospital days
  The EuroQol EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. The EuroQol visual analogue scale (EQ VAS) records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. Detailed scoring instructions are available: https://euroqol.org/wp-content/uploads/2016/09/EQ-5D-3L_UserGuide_2015.pdf

OTHER OUTCOMES:
Pain Treatment Satisfaction Scale | Assessed once at the end of hospital stay (average length of stay = 5 days)
  The Pain Treatment Satisfaction Scale includes subscales of satisfaction with information, medical care, effectiveness, and side effects with reliability ranging from 0.83 to 0.92. Each of the subscales are scored from 0 to 100 with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Chao, DrPH, MPA, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No